CLINICAL TRIAL: NCT05961839
Title: A First-In-Human, Phase 1, Dose Escalation Study of SGR-2921 as Monotherapy In Subjects With Relapsed/Refractory Acute Myeloid Leukemia or Myelodysplastic Syndrome
Brief Title: Study of SGR-2921 in Relapsed/Refractory Acute Myeloid Leukemia or Myelodysplastic Syndrome
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company decision
Sponsor: Schrödinger, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SGR-2921-101
Record Dates: First submitted 2023-07-17; First posted 2023-07-27 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia; High-Risk and Very High-Risk Myelodysplastic Syndromes
Keywords: MDS; Relapsed or Refractory AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation in the Absence of Specific Azole Antifungal Treatments (Experimental): Up to 9 dose levels will be evaluated in subjects not receiving specific azole antifungal treatment.
  Interventions: Drug: SGR-2921
- Dose Escalation in the Presence of Specific Azole Antifungal Treatments (Experimental): Up to 9 dose levels will be evaluated in subjects receiving specific azole antifungal treatment.
  Interventions: Drug: SGR-2921

INTERVENTIONS:
Drug: SGR-2921 — SGR-2921 will be administered orally.

SUMMARY:
The purpose of this study is to evaluate safety and tolerability and to determine the maximum tolerated dose (MTD) and/or recommended dose (RD) of SGR-2921.

DETAILED DESCRIPTION:
This is a study of SGR-2921, an oral, small molecule inhibitor of cell division cycle 7-related protein kinase (CDC7), in subjects with Relapsed/Refractory (R/R) Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS) to evaluate the safety, pharmacokinetics (PK), pharmacodynamics (PD), maximum tolerated dose (MTD) and/or recommended dose (RD) of SGR-2921.

Exploratory cohorts may evaluate additional PK, PD, preliminary anti-tumor activity, and safety to establish the SGR-2921 RD. A planned amendment will evaluate SGR-2921 in combination with other approved AML/MDS treatments such as hypomethylating agents (HMA), BCL2 inhibitors, IDH inhibitors or FLT3 inhibitors, in patients with AML and/or MDS.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age.
* Life expectancy ≥ 8 weeks.
* Confirmed diagnosis of R/R AML or High Risk (HR) and Very High Risk (VHR) MDS.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.

Exclusion Criteria:

* Active malignancies within two years prior to the first dose, or requiring ongoing treatment, not related to AML or MDS.
* Clinical evidence of central nervous system (CNS) or pulmonary leukostasis, ≥ Grade 3 disseminated intravascular coagulation, or active CNS leukemia.
* Use of experimental drug, or therapy, or anti-cancer therapy within 14 days or 5 half-lives of the first dose of study drug.
* QT interval corrected for heart rate per Fridericia's formula ≥470 msec during screening ECG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities | From first dose until the end of Cycle 1 (approximately 28 days, up to 42 days).
Adverse Events | Throughout the study, up to 26 months.
  Incidence, nature, and severity of adverse events (AEs) as assessed by the NCI CTCAE v5.0.
Electrocardiograms in Singlicate and Triplicate | Throughout the study, up to 26 months.
  Uncorrected QT interval, QTcF, PR duration, QRS interval, and RR interval.

SECONDARY OUTCOMES:
SGR-2921 Maximal Plasma Concentration (Cmax) | Throughout the study, up to 26 months.
  Concentrations of SGR-2921 in plasma are measured at various timepoints following its administration to calculate typical exposure/PK parameters, including, but not limited to, the maximal plasma concentration (Cmax).
SGR-2921 Minimum Plasma Concentration (Cmin) | Throughout the study, up to 26 months.
  Concentrations of SGR-2921 in plasma are measured at various timepoints following its administration to calculate typical exposure/PK parameters, including, but not limited to, the minimum plasma concentration (Cmin).
SGR-2921 Time to Maximal Plasma Concentration (tmax) | Throughout the study, up to 26 months.
  Concentrations of SGR-2921 in plasma are measured at various timepoints following its administration to calculate typical exposure/PK parameters, including, but not limited to, the time to maximal plasma concentration (tmax).
SGR-2921 Area Under the Concentration Versus Time Curve (AUC) | Throughout the study, up to 26 months.
  Concentrations of SGR-2921 in plasma are measured at various timepoints following its administration to calculate typical exposure/PK parameters, including, but not limited to, the area under the concentration versus time curve (AUC).
Composite Complete Remission (CR) Rate for Subjects with AML | Throughout the study, up to 26 months.
  The percentage of subjects with CR, CR with Partial Hematologic Recovery (CRh), and CR with Incomplete Blood Count Recovery (CRi).
Objective Response Rate (ORR) for Subjects with AML | Throughout the study, up to 26 months.
  The percentage of subjects achieving CR, CRh, CRi, morphologic leukemia-free state (MLFS) and Partial Response (PR).
Objective Response Rate (ORR) for Subjects with MDS | Throughout the study, up to 26 months.
  The percentage of subjects achieving CR and PR.
Duration of Response (DOR) for Subjects with AML | Throughout the study, up to 26 months.
  The time from first response (CR, CRh, CRi, MLFS, or PR) to the date of initial objectively documented progression or death due to any cause, whichever occurs first.
Duration of Response (DOR) for subjects with MDS | Throughout the study, up to 26 months.
  The time from first response (CR or PR) to the date of initial objectively documented progression or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Weiss, M.D., Study Director — Schrödinger, Inc.
Locations (12):
- United States (12):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - The University of Kansas Clinical Research Center, Fairway, Kansas
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center - James Cancer Hospital, Columbus, Ohio
  - Oncology Associates of Oregon, P.C., Eugene, Oregon
  - Oregon Health & Science University - Knight Cancer Institute - Center of Hematologic Malignancies, Portland, Oregon
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Clinical Research Organization, Philadelphia, Pennsylvania
  - TriStar Bone Marrow Transplant, LLC, Nashville, Tennessee
  - St. David's South Austin Medical Center, Austin, Texas
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No